CLINICAL TRIAL: NCT05746520
Title: Complex And Simple Appendicitis: REstrictive or Liberal Post-operative Antibiotic eXposure (CASA RELAX) Using Desirability of Outcome Ranking (DOOR) and Response Adjusted for Duration of Antibiotic Risk (RADAR)
Brief Title: Complex And Simple Appendicitis: REstrictive or Liberal Post-operative Antibiotic eXposure (CASA RELAX) - Atrium Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00086118
Record Dates: First submitted 2023-02-16; First posted 2023-02-27 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-01

CONDITIONS: Appendicitis Surgery
Keywords: post-operative antibiotics; acute appendicitis; complicated appendicitis
MeSH Terms: conditions — Appendicitis | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Restricted Post-Operative Antibiotics Group (Experimental): Participants undergoing standard of care (SOC) with simple appendicitis will not receive post-operative antibiotics.
  Participants undergoing standard of care (SOC) with complicated (gangrenous or perforated) appendicitis will receive 24 hours of SOC post-operative antibiotics.
  Interventions: Other: Antibiotic
- Restricted Duration of SOC Antibiotic Use (Other): Use of Standard of Care Antibiotics, type as determined by the clinician, will be restricted to none or 24 hours of post-operatively.
  Interventions: Other: Antibiotic
- Liberal Post-Operative Antibiotics Group (Active Comparator): Participants undergoing standard of care (SOC) with simple appendicitis will receive 24 hours of post-operative antibiotics.
  Participants undergoing standard of care (SOC) with complicated (gangrenous or perforated) appendicitis will receive 4 days of SOC post-operative antibiotics.
  Interventions: Other: Antibiotic
- Liberal Duration of SOC Antibiotic Use (Other): Use of Standard of Care Antibiotics, type as determined by the clinician, will be permitted for 24 hours or 4 days of post-operatively.
  Interventions: Other: Antibiotic

INTERVENTIONS:
Other: Antibiotic — Type of antibiotic is per clinical judgement with the duration being the experimental aspect of this study.
  Other Names: antibiotics are per standard of care (SOC)

SUMMARY:
To demonstrate the safety, efficacy, and feasibility of short-course post-operative antibiotic treatment for simple and complicated appendicitis

DETAILED DESCRIPTION:
This is a single center, randomized controlled trial to determine if decreasing the amount of antibiotics after appendicitis surgery can decrease the risk of adverse effects associated with antibiotics while at the same time ensuring participant safety.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Planned appendectomy (laparoscopic or open)
* Willing and able to provide informed consent
* Working telephone number or reliable method to contact patient after hospital discharge

Exclusion Criteria:

* Unable to consent
* Pregnant Women
* Prisoners
* immunocompromised as determined by clinical team, or patients actively receiving steroids, chemotherapy, or immunosuppressing medications (for example tacrolimus), or patients with active hematologic malignancy affecting the immune system, leukopenia, or end-stage Acquired immunodeficiency syndrome (AIDS)
* Heart Failure
* Allergy to Bupivacaine
* Unlikely to comply with treatment or follow-up
* Inpatient consultation for appendicitis
* Clinically suspected sepsis based on Sepsis-3 definition
* Current use of antibiotics for other indications
* Type 1 Diabetes or uncontrolled hyperglycemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2023-03-02 (Actual); Primary Completion 2025-06-18 (Actual); Study Completion 2025-07-21 (Actual)

PRIMARY OUTCOMES:
Number of participants with no antibiotic related adverse effects | Day 30
  All subjects will be contacted at least 30 days after appendectomy by telephone if unable to contact subject, then electronic medical record will be reviewed. Outcomes will be assessed by Desirability of Outcome Ranking (DOOR), with the lowest ranking of 1 indicating no adverse effects. Infectious/antibiotic complications requiring antibiotic treatment only, Emergency Department visit, hospital readmission, percutaneous drainage, operative intervention, and death ranked 2 through 7. A lower score indicates a more desirable outcome. For subjects of same DOOR score, Response Adjusted for Duration of Antibiotic Risk (RADAR) scores will be used to determine the better outcome. The distribution of DOOR scores and associated statistical analyses will be reported.

SECONDARY OUTCOMES:
Incidence of Infectious/Antibiotic Complications | Day 30
  All subjects will be monitored from consent until follow up at least 30 days after appendectomy for number of complications. Each event will be assessed by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v.5.0, with the lowest grade being 1 and the highest grade of 5 indicating death. A higher grade indicates a more serious event.

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Torres Fajardo, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
de-identified data will be shared with Denver health and combined with data from other independent sites for final analysis
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose

DOCUMENTS (1):
  • Informed Consent Form (2025-06-27): https://cdn.clinicaltrials.gov/large-docs/20/NCT05746520/ICF_000.pdf